CLINICAL TRIAL: NCT02126592
Title: The Secretion of Incretin Hormones in Patients With Polycystic Ovary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 12XJ10015
Record Dates: First submitted 2014-01-21; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-01

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — only plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PCOS cohort: Women with PCOS
- Control cohort: Women without PCOS

SUMMARY:
Polycystic ovary syndrome (PCOS) is an endocrine disease in reproductive women. It is characterized by anovulation and hyperandrogenism. Most patients with PCOS have metabolic abnormalities such as dyslipidemia, insulin resistance and glucose abnormalities. Almost 60-80﹪PCOS patients are obesity which exacerbates IR and hyperandrogenism. Obese PCOS patients tend to be overeating suggests that impaired appetite regulation might be contribute to the pathophysiology of PCOS. Our study is trying to observe difference of incretin between PCOS and normal control to figure out whether change of incretin is involved in the pathophysiology of PCOS.

ELIGIBILITY:
Inclusion Criteria:

* women at reproductive age
* women with PCOS and women without PCOS

Exclusion Criteria:

* young women who had their menarche less than 3 years
* women older than 45 years old, Amenorrhea of menopause, hyperglycemia, hyperthyroidism, hypothyroidism, heart failure, lung failure, renal failure, anemia, dystrophy, gonitis

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Polycystic Ovary Syndrome(PCOS)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-04 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Change in incretin hormones secretion in PCOS patients. | up to 14 months

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, China